CLINICAL TRIAL: NCT01022099
Title: Prospective Randomized Trial of Navigated and Conventional TKA With Radiographic and CT Evaluations
Brief Title: Prospective Randomized Trial of Navigated and Conventional TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Dresden University of Technology, Dr Joerg Luetzner, Dresden University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KneeNavy
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Total Knee Arthroplasty; Navigation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- navigated TKA (Active Comparator)
  Interventions: Procedure: Implantation of a Total Knee Arthroplasty
- conventional TKA (Other)
  Interventions: Procedure: Implantation of a Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Implantation of a Total Knee Arthroplasty — In all patients a cemented, unconstrained, cruciate-retaining TKA with a rotating platform (ScorpioTM PCS, Stryker Orthopaedics, Mahwah, NJ) was implanted. No patellar resurfacing was performed. A medial parapatellar approach with a femur-first preparation was done in all cases.
  The Stryker Navigation System, Knee Navigation Software V3.1 (Stryker Orthopaedics, Mahwah, NJ) was used for computer-assisted implantation.
  The conventional implantation was performed with femoral intramedullary and tibial extramedullary standard alignment guides.
  Other Names: ScorpioTM PCS; Stryker Navigation System; Stryker Knee Navigation Software V3.1

SUMMARY:
Evaluation of the component position and kinematics after navigated and conventional Total Knee Arthroplasty.

DETAILED DESCRIPTION:
1. Component position, kinematics After skin closure lateral x-rays were done in different flexion angles in order to evaluate the kinematic behaviour of the TKA.

   A full-length standing and a lateral radiograph as well as CT scans of the hip, knee and ankle joint were performed 5 to 7 days postoperatively before discharge.
2. clinical outcome Patient sociodemographic and anamnestic data were collected. The written interview was complemented by the EuroQol questionnaire (release EQ-5D) and the assessment of the patients' functional status (Knee Society Score) one week before surgery and 18 to 24 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary osteoarthritis of the knee
* indication to TKA
* a mechanical axis between 20° varus and 5° valgus
* signed informed consent

Exclusion Criteria:

* previous hemi- or total arthroplasty
* severe instability that could not be treated with an unconstrained, cruciate-retaining TKA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
rotational component position | postoperatively

SECONDARY OUTCOMES:
leg axis | postoperatively
kinematics | postoperatively
clinical outcome | 18 to 24 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Peter Günther, MD, PhD, Study Director — Orthopaedic Department, University Hospital Dresden
Locations (1):
- University Hospital Dresden, Orthopaedic Department, Dresden, Germany

REFERENCES:
- [Result] Lutzner J, Krummenauer F, Wolf C, Gunther KP, Kirschner S. Computer-assisted and conventional total knee replacement: a comparative, prospective, randomised study with radiological and CT evaluation. J Bone Joint Surg Br. 2008 Aug;90(8):1039-44. doi: 10.1302/0301-620X.90B8.20553. PMID 18669959
- [Derived] Beyer F, Pape A, Lutzner C, Kirschner S, Lutzner J. Similar outcomes in computer-assisted and conventional total knee arthroplasty: ten-year results of a prospective randomized study. BMC Musculoskelet Disord. 2021 Aug 18;22(1):707. doi: 10.1186/s12891-021-04556-3. PMID 34407776
- [Derived] Harman MK, Banks SA, Kirschner S, Lutzner J. Prosthesis alignment affects axial rotation motion after total knee replacement: a prospective in vivo study combining computed tomography and fluoroscopic evaluations. BMC Musculoskelet Disord. 2012 Oct 23;13:206. doi: 10.1186/1471-2474-13-206. PMID 23088451
- [Derived] Lutzner J, Krummenauer F, Gunther KP, Kirschner S. Rotational alignment of the tibial component in total knee arthroplasty is better at the medial third of tibial tuberosity than at the medial border. BMC Musculoskelet Disord. 2010 Mar 25;11:57. doi: 10.1186/1471-2474-11-57. PMID 20338042